CLINICAL TRIAL: NCT05564572
Title: Randomized Implementation of Routine Patient-Reported Health Status Assessment Among Heart Failure Patients in Stanford Cardiology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alexander Sandhu, Instructor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 67173
Record Dates: First submitted 2022-09-01; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Status Assessment (Experimental): Completion of a patient-reported health status assessment preceding each clinic visit. The health status assessment consists of the Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) along with additional select questions. The results of the assessment will be available to clinicians in the electronic health record.
  Interventions: Other: Routine Health Status Assessment
- Usual Care (No Intervention): Patients will not complete a patient-reported health status measures.

INTERVENTIONS:
Other: Routine Health Status Assessment — Completion of a patient-reported health status assessment preceding each clinic visit. The health status assessment consists of the Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) along with additional select questions. The results of the assessment will be available to clinicians in the electronic health record.
  Arms: Health Status Assessment

SUMMARY:
This randomized quality improvement study evaluates the routine assessment of patient-reported heath status, using the Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) among adult outpatients seen in heart failure clinic or seen in general cardiology clinic with a history of heart failure. Patients will be randomized 4:1 to KCCQ-12 assessment or usual care. Participants randomized to KCCQ-12 assessment will complete the KCCQ-12 at every heart failure clinic visit. Their results will be available to clinicians to assist with clinical management. Heath status surveys will not be integrated into clinical care for patients in the usual care arm. The primary objective is to evaluate the impact of routine assessment of patient-reported heath status on clinical processes of care. As the primary outcome, we will evaluate clinician inertia by measuring the clinician action rating (CAR) - an aggregate count of medication changes, referrals, and diagnostic tests. As secondary outcomes, we will measure individual components of the composite outcome, therapy rates, resource utilization, and patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Seen in Stanford general cardiology clinic with a diagnosis of heart failure or cardiomyopathy or in heart failure clinic

Exclusion Criteria:

* Enrolled in PRO-HF trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-09-07 (Estimated); Study Completion 2023-12-07 (Estimated)

PRIMARY OUTCOMES:
Clinician action rating | From date of randomization to study completion (up to 12 months)
  Aggregate count of medication changes, referrals, and diagnostic tests ordered per clinic visit

SECONDARY OUTCOMES:
Medication Changes | From date of randomization to study completion (up to 12 months)
  Number of medication changes per cardiology clinic visit (initiation, discontinuation, dose adjustment)
Referrals | From date of randomization to study completion (up to 12 months)
  Number of referrals per cardiology clinic visit
Diagnostic Tests | From date of randomization to study completion (up to 12 months)
  Number of diagnostic tests ordered per cardiology clinic visit
Percentage of Patients on Beta-blocker Therapy and Median Dose Among Patients with Reduced Ejection Fraction | From date of randomization to study completion (up to 12 months)
  Beta-blocker therapy use among the sub-group of patients with baseline left ventricular ejection fraction ≤ 40%. Among those patients on therapy, the specific medication and dose will be collected.
Percentage of Patients on Renin-Angiotensin-Aldosterone System Inhibitors and Median Dose Among Patients with Reduced Ejection Fraction | From date of randomization to study completion (up to 12 months)
  Use of any renin-angiotensin-aldosterone system inhibitors among the sub-group of patients with baseline left ventricular ejection fraction ≤ 40%. These include angiotensin-converting enzyme inhibitor, angiotensin receptor blockers, or angiotensin receptor-neprilysin inhibitors. Among those patients on therapy, the specific medication and dose will be collected.
Percentage of Patients on Mineralocorticoid Receptor Antagonist and Median Dose Among Patients with Reduced Ejection Fraction | From date of randomization to study completion (up to 12 months)
  Mineralocorticoid receptor antagonist use among the sub-group of patients with baseline left ventricular ejection fraction ≤ 40%. Among those patients on therapy, the specific medication and dose will be collected.Mineralocorticoid receptor antagonist use among the sub-group of patients with left ventricular ejection fraction ≤ 40%. Among those patients on therapy, the specific medication and dose will be collected.
  Mineralocorticoid receptor antagonist use among the sub-group of patients with left ventricular ejection fraction ≤ 40%. Among those patients on therapy, the specific medication and dose will be collected.
Percentage of Patients on Sacubitril-Valsartan and Median Dose Among Patients with Reduced Ejection Fraction | From date of randomization to study completion (up to 12 months)
  Use of any sacubitril-valsartan among the sub-group of patients with baseline left ventricular ejection fraction ≤ 40%. These include angiotensin-converting enzyme inhibitor, angiotensin receptor blockers, or angiotensin receptor-neprilysin inhibitors. Among those patients on therapy, the specific medication and dose will be collected.
Percentage of Patients on SGLT2i | From date of randomization to study completion (up to 12 months)
  Use of any SGLT2i
Percentage of Patients with a Implantable Cardiac Defibrillator Among Patients with Reduced Ejection Fraction | From date of randomization to study completion (up to 12 months)
  Presence of an implantable cardiac defibrillator among the sub-group of patients with baseline left ventricular ejection fraction ≤ 35%.
Percentage of Patients with a Cardiac Resynchronization Therapy Device Among Patients with Reduced Ejection | From date of randomization to study completion (up to 12 months)
  Presence of cardiac resynchronization therapy among the sub-group of patients with baseline left ventricular ejection fraction ≤ 35% with electrocardiogram findings consistent with the guideline recommendation for cardiac resynchronization therapy.
Percentage of Patients Given Cardiac Rehabilitation Referral Among Patients with Reduced Ejection Fraction | From date of randomization to study completion (up to 12 months)
  Referral to cardiac rehabilitation among the subgroup of patients with baseline left ventricular ejection fraction ≤ 35%.
Hospitalizations | From date of randomization to study completion (up to 12 months)
  Number of heart failure hospitalizations and non-heart failure hospitalizations in the Stanford healthcare system during the follow-up period.
Emergency Department Visits | From date of randomization to study completion (up to 12 months)
  Number of Stanford emergency department visits during the follow-up period
Cardiology Clinic Visits | From date of randomization to study completion (up to 12 months)
  Number of visits (in-person or telemedicine) to general cardiology or heart failure clinics during the follow-up period
Telephone Encounters | From date of randomization to study completion (up to 12 months)
  Number of telephone encounters with general cardiology or heart failure clinics during the follow-up period
Formal Advanced Heart Failure Therapy Evaluation | From date of randomization to study completion (up to 12 months)
  Number of patients who undergo formal evaluation for advanced heart failure therapies (LVAD or transplant)
Quality of Patient Clinic Experience | From date of randomization to study completion (up to 12 months)
  Patient report of satisfaction with clinic visit based on existing Stanford patient experience survey
Diagnostic Testing | From date of randomization to study completion (up to 12 months)
  Number of diagnostic tests ordered in cardiology clinic (cardiac imaging [echocardiography, MRI, angiography, CT angiography, PET], non-cardiac imaging, rhythm monitoring, exercise testing, invasive hemodynamics, pulmonary function testing) during the follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Hospital & Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No